CLINICAL TRIAL: NCT06562101
Title: Effects of Intra-articular Stromal Vascular Fraction Injection on Clinical Symptoms and Cartilage Health in Osteoarthritic Knees: A Single-Center Pilot Study
Brief Title: Effects of Intra-articular Stromal Vascular Fraction Injection on Clinical Symptoms and Cartilage Health in Osteoarthritic Knees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shu-Hao Chang, MD (Other)
Responsible Party: Sponsor-Investigator, Shu-Hao Chang, MD, Visiting staff, Fu Jen Catholic University Hospital
Organization: Fu Jen Catholic University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FJUH109069
Record Dates: First submitted 2024-08-14; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stromal Vascular Fraction (SVF) (Experimental): Ten patients with knee OA were administered intra-articular SVF injections.
  Interventions: Procedure: Intra-articular Stromal Vascular Fraction Injection

INTERVENTIONS:
Procedure: Intra-articular Stromal Vascular Fraction Injection — Adipose tissue was harvested using the Q-graft system (Human Med®) from the abdominal subcutaneous fat of patients under local anesthesia. After concentration and resuspension in normal saline, 5 mL of the SVF suspension was injected into the knee joint cavity under sterile conditions.
  Other Names: Stromal Vascular Fraction therapy

SUMMARY:
Background: Osteoarthritis (OA) is a prevalent form of arthritis worldwide. Intra-articular stromal vascular fraction (SVF) injections are a potential therapeutic option for patients with OA. This study aims to assess the effects of intra-articular SVF injections on knee OA. Methods: Ten patients with knee OA participated in this study. After being administered intra-articular SVF injections, their outcomes were evaluated using various questionnaires. MRI T2 mapping was conducted and compared before the intervention and 6 months after. All data underwent analysis using various tests.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 35 years.
* Patients with degenerative knee OA confirmed via X-ray and classified according to the Kellgren Lawrence Grading Scale 2~4.
* Persistent knee pain after nonsurgical treatment.

Exclusion Criteria:

* Arthritis caused by other systemic or local immune diseases.
* Patients who have undergone total knee replacement surgery.
* Patients who have been administered platelet-rich plasma or hyaluronic acid injections within the past three months.
* Patients with symptoms related to degenerative arthritis in the ankle, which affected the assessment of pain.
* Patients with severe heart problems and coagulation disorders.
* Patients who have taken glucosamine within the previous month.
* MRI exclusion conditions, including patients with a heart rhythm regulator who have received vascular surgery with a hemostatic clip and artificial heart valves.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline and at 3 and 6 months post-intervention
  range from 0-96, with higher scores indicating greater OA-related disability
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline and at 3 and 6 months post-intervention
  5 items, ranging from 0-96, with higher scores indicating worse life quality related to OA
Visual Analogue Scale (VAS) | Baseline and at 3 and 6 months post-intervention
  range from 0-10, with higher scores indicating increased degree of pain
Magnetic resonance imaging (MRI) | Baseline and 6 months after the intervention
  included T2 mapping

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Hao Chang, MD, Principal Investigator — Department of Orthopedics, Fu Jen Catholic University Hospital, Fu Jen Catholic University
Locations (1):
- Fu Jen Catholic University Hospital, New Taipei City, Taiwan

REFERENCES:
- [Background] Abramoff B, Caldera FE. Osteoarthritis: Pathology, Diagnosis, and Treatment Options. Med Clin North Am. 2020 Mar;104(2):293-311. doi: 10.1016/j.mcna.2019.10.007. Epub 2019 Dec 18. PMID 32035570
- [Background] Lin FH, Chen HC, Lin C, Chiu YL, Lee HS, Chang H, Huang GS, Chang HL, Yeh SJ, Su W, Wang CC, Su SL. The increase in total knee replacement surgery in Taiwan: A 15-year retrospective study. Medicine (Baltimore). 2018 Aug;97(31):e11749. doi: 10.1097/MD.0000000000011749. PMID 30075592
- [Background] Taruc-Uy RL, Lynch SA. Diagnosis and treatment of osteoarthritis. Prim Care. 2013 Dec;40(4):821-36, vii. doi: 10.1016/j.pop.2013.08.003. Epub 2013 Sep 26. PMID 24209720
- [Background] Garza JR, Campbell RE, Tjoumakaris FP, Freedman KB, Miller LS, Santa Maria D, Tucker BS. Clinical Efficacy of Intra-articular Mesenchymal Stromal Cells for the Treatment of Knee Osteoarthritis: A Double-Blinded Prospective Randomized Controlled Clinical Trial. Am J Sports Med. 2020 Mar;48(3):588-598. doi: 10.1177/0363546519899923. PMID 32109160
- [Background] Coughlin RP, Oldweiler A, Mickelson DT, Moorman CT 3rd. Adipose-Derived Stem Cell Transplant Technique for Degenerative Joint Disease. Arthrosc Tech. 2017 Oct 2;6(5):e1761-e1766. doi: 10.1016/j.eats.2017.06.048. eCollection 2017 Oct. PMID 29399463
- [Background] Lamo-Espinosa JM, Mora G, Blanco JF, Granero-Molto F, Nunez-Cordoba JM, Sanchez-Echenique C, Bondia JM, Aquerreta JD, Andreu EJ, Ornilla E, Villaron EM, Valenti-Azcarate A, Sanchez-Guijo F, Del Canizo MC, Valenti-Nin JR, Prosper F. Intra-articular injection of two different doses of autologous bone marrow mesenchymal stem cells versus hyaluronic acid in the treatment of knee osteoarthritis: multicenter randomized controlled clinical trial (phase I/II). J Transl Med. 2016 Aug 26;14(1):246. doi: 10.1186/s12967-016-0998-2. PMID 27565858
- [Background] Lindroos B, Suuronen R, Miettinen S. The potential of adipose stem cells in regenerative medicine. Stem Cell Rev Rep. 2011 Jun;7(2):269-91. doi: 10.1007/s12015-010-9193-7. PMID 20853072
- [Background] Dahaghin S, Bierma-Zeinstra SM, Ginai AZ, Pols HA, Hazes JM, Koes BW. Prevalence and pattern of radiographic hand osteoarthritis and association with pain and disability (the Rotterdam study). Ann Rheum Dis. 2005 May;64(5):682-7. doi: 10.1136/ard.2004.023564. Epub 2004 Sep 16. PMID 15374852
- [Background] Dillon CF, Rasch EK, Gu Q, Hirsch R. Prevalence of knee osteoarthritis in the United States: arthritis data from the Third National Health and Nutrition Examination Survey 1991-94. J Rheumatol. 2006 Nov;33(11):2271-9. Epub 2006 Oct 1. PMID 17013996
- [Background] Xia B, Di Chen, Zhang J, Hu S, Jin H, Tong P. Osteoarthritis pathogenesis: a review of molecular mechanisms. Calcif Tissue Int. 2014 Dec;95(6):495-505. doi: 10.1007/s00223-014-9917-9. Epub 2014 Oct 14. PMID 25311420
- [Background] Krasnokutsky S, Samuels J, Abramson SB. Osteoarthritis in 2007. Bull NYU Hosp Jt Dis. 2007;65(3):222-8. PMID 17922674
- [Background] Anil U, Markus DH, Hurley ET, Manjunath AK, Alaia MJ, Campbell KA, Jazrawi LM, Strauss EJ. The efficacy of intra-articular injections in the treatment of knee osteoarthritis: A network meta-analysis of randomized controlled trials. Knee. 2021 Oct;32:173-182. doi: 10.1016/j.knee.2021.08.008. Epub 2021 Sep 6. PMID 34500430
- [Background] Aletto C, Giordano L, Quaranta M, Zara A, Notarfrancesco D, Maffulli N. Short-term results of intra-articular injections of stromal vascular fraction for early knee osteoarthritis. J Orthop Surg Res. 2022 Jun 11;17(1):310. doi: 10.1186/s13018-022-03196-0. PMID 35690837
- [Background] Friedrich KM, Shepard T, de Oliveira VS, Wang L, Babb JS, Schweitzer M, Regatte R. T2 measurements of cartilage in osteoarthritis patients with meniscal tears. AJR Am J Roentgenol. 2009 Nov;193(5):W411-5. doi: 10.2214/AJR.08.2256. PMID 19843720
- [Background] Zhang Y, Bi Q, Luo J, Tong Y, Yu T, Zhang Q. The Effect of Autologous Adipose-Derived Stromal Vascular Fractions on Cartilage Regeneration Was Quantitatively Evaluated Based on the 3D-FS-SPGR Sequence: A Clinical Trial Study. Biomed Res Int. 2022 Jan 25;2022:2777568. doi: 10.1155/2022/2777568. eCollection 2022. PMID 35118156